CLINICAL TRIAL: NCT05885451
Title: A Phase I, Double Blind, Placebo-controlled, Randomized, Parallel, Single Ascending Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of AMG 592 Administered Subcutaneously in Healthy Japanese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of AMG 592 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20180132
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-04

CONDITIONS: Chronic Graft-versus-Host Disease (cGVHD)
Keywords: Chronic Graft-versus-Host Disease; AMG 592; Inflammatory Conditions
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: AMG 592 Dose 1 (Experimental): Participants will receive AMG 592 dose 1 subcutaneously
  Interventions: Drug: AMG 592
- Arm 2: AMG 592 Dose 2 (Experimental): Participants will receive AMG 592 dose 2 subcutaneously
  Interventions: Drug: AMG 592
- Arm 3: Placebo (Placebo Comparator): Participants will receive placebo subcutaneously
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMG 592 — Administered as SC injection
  Arms: Arm 1: AMG 592 Dose 1; Arm 2: AMG 592 Dose 2
Other: Placebo — Administered as SC injection
  Arms: Arm 3: Placebo

SUMMARY:
The primary objective of this study is to characterize the pharmacokinetics (PK) profile of a single dose of AMG 592 administered subcutaneously in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be first generation Japanese (4 grandparents, biologic parents, and subject born in Japan and of Japanese heritage)
* Male and female participants must be ≥ 18 and ≤ 55 years of age with a body mass index (BMI) of ≥ 18.5 and ≤ 25.0 kg/m^2 at the time of screening

Exclusion Criteria:

* Participant with history of prior malignancy within the last 5 years except malignancy (in situ) fully excised or treated with curative intent and with no known active disease present for ≥3 years before enrollment and felt to be at low risk for recurrence by the treating physician, non-melanoma skin cancers, cervical or breast ductal carcinoma in situ
* Participants with a known history of autoimmune disease
* Participants who have donated or lost ≥ 500 mL of blood or plasma within 8 weeks of administration of the first dose of IP
* Participants with any active infection for which systemic anti-infectives were used within 4 weeks prior to Day 1
* Positive for Hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B)
* Participant has positive test results for Human Immunodeficiency Virus (HIV)
* Participant has a positive test for tuberculosis during screening defined as either a positive purified derivative (PPD) (>= 5 mm of induration at 48 to 72 hours after test is placed) OR a positive QuantiFERON test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of AMG 592 | Up to Day 43
Time of Maximum Observed Concentration (tmax) of AMG 592 | Up to Day 43
Area Under the Serum Concentration-time Curve to the Last Measurable Point (AUClast) of AMG 592 | Up to Day 43
Area Under the Concentration-time Curve (AUC) from Time Zero to Infinity (AUCinf) | Up to Day 43

SECONDARY OUTCOMES:
Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) | Day 1 to Day 43
Number of Participants who Experience Anti-AMG 592 Antibodies Formation | Up to Day 43

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com